CLINICAL TRIAL: NCT02729285
Title: Preoperative Ketorolac for Intraoperative and Postoperative Pain Management in Scleral Buckling Surgery Under Retrobulbar Block Anesthesia: A Prospective, Randomized, Controlled Study
Brief Title: Preoperative Ketorolac for Pain Control in Scleral Buckle Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Lu, Director, Fundus Disease Center of Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2014MEKY042
Record Dates: First submitted 2016-03-27; First posted 2016-04-06 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ketorolac Tromethamine; Ketorolac; Scleral Buckling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketorolac Tromethamine (Experimental): On operation day, the patients were randomly assigned to receive intramuscular Ketorolac 60-mg 30 minutes before scleral buckle surgery.
  Interventions: Drug: Ketorolac Tromethamine; Procedure: scleral buckle
- placebo (Placebo Comparator): On operation day, the patients were randomly assigned to receive placebo before scleral buckle surgery.
  Interventions: Drug: placebo; Procedure: scleral buckle

INTERVENTIONS:
Drug: Ketorolac Tromethamine — On operation day, the patients were randomly assigned to receive intramuscular Ketorolac 60-mg 30 min before scleral buckle surgery.
  Other Names: ketorolac
  Arms: Ketorolac Tromethamine
Drug: placebo — On operation day, the patients were randomly assigned to receive placebo 30 min before scleral buckle surgery.
  Other Names: disambiguation
  Arms: placebo
Procedure: scleral buckle — Surgical procedure of scleral buckle under retrobulbar block anesthesia

SUMMARY:
The scleral buckle surgery is an effective way in treating retinal detachment (RD) patients. Retrobulbar block has been proved effective in scleral buckle surgery. Though retrobulbar anesthesia saves operative time and money compared to general analgesia, the intraoperative pain is frequent and a proportion of postoperative pain is often ignored. Ketorolac has been demonstrated to be a preemptive analgesia in other diseases such as adenotonsillectomy, posterior lumbar spinal fusion, laser-assisted subepithelial keratectomy (LASEK), and so forth. The aim of the investigators study is to determine the safety and preemptive analgesic effect of ketorolac in the perioperative pain control of patients undergoing RD surgery under retrobulbar anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. consent of the patient or legal guardian
2. 18 years or above
3. normal height and weight
4. ASA class I, II
5. elective surgery
6. surgery time within 60min
7. understanding of the verbal numerical rating score (0-10)

Exclusion Criteria:

1. history of ocular surgery, trauma or infection
2. intraoperative complications
3. glaucoma or ocular hypertension (> 20 mmHg)
4. diabetic retinopathy
5. diagnosis of asthma or coagulopathy
6. chronic pain syndromes
7. history of peptic ulceration, liver or hematologic disease
8. history of chronic use of analgesics, sedatives, opioids or steroids
9. history of drug or alcohol abuse
10. history of systemic disease
11. sexually transmitted disease (STD)
12. Pregnancy, lactation;
13. cognitive impairment or psychiatric illness;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pain score using numerical rating scale (NRS) | preoperative
Pain score using numerical rating scale (NRS) | intraoperative
  any pain during the whole operation time
Pain score using numerical rating scale (NRS) | immediately after operation
Pain score using numerical rating scale (NRS) | at 4 hours postoperatively
Pain score using numerical rating scale (NRS) | at 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Lu Lin, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen X, Liu B, Liang X, Li J, Li T, Li Y, Yu X, Lyu C, Zhao X, Tanumiharjo S, Jin C, Lu L. The Combination of Ketorolac with Local Anesthesia for Pain Control in Day Care Retinal Detachment Surgery: A Randomized Controlled Trial. J Ophthalmol. 2017;2017:3464693. doi: 10.1155/2017/3464693. Epub 2017 Jul 9. PMID 28770108